CLINICAL TRIAL: NCT02209597
Title: Bioequivalence and Clinical Effects of Generic and Brand Bupropion
Brief Title: Clinical Study of Generic and Brand Bupropion in Depression
Acronym: BALANCE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 201312021
Record Dates: First submitted 2014-07-07; First posted 2014-08-06 (Estimated); Results first posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; bupropion XL; Wellbutrin XL
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Bupropion; Pregnane X Receptor

STUDY DESIGN:
Intervention Model Description: Each participant receives the 4 drugs in sequence (sequence is randomized).
Who Masked: Participant, Care Provider
Masking Description: The randomization table will be generated by the Barnes-Jewish Hospital Investigational Pharmacy. Each subject will be assigned the next available number. Subjects, investigators, and all study team members will be blinded to drug treatment. In the case of dropouts (either subject- or investigator-initiated), subjects will be replaced, to provide the required number of subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- StudyArm (Experimental): Subjects will be studied for 28 weeks in a sequential cross-over study: a
  Subjects will be studied in 4 phases for a total of approximately 28 weeks:
  Phase 1: an approximately 4-week lead-in phase during which participants remain on their existing bupropion product Phases 2 - 4: randomized cross-over phases of approximately 6 weeks on each of the four bupropion study drugs (brand and 3 generics).
  Interventions: Drug: Bupropion XL 300

INTERVENTIONS:
Drug: Bupropion XL 300 — Subjects will be studied in 4 phases for a total of approximately 28 weeks:
  Phase 1: an approximately 4-week lead-in phase during which participants remain on their existing bupropion product Phases 2 - 4: randomized cross-over phases of approximately 6 weeks on each of the four bupropion study drugs (brand and 3 generics).
  Other Names: Wellbutrin; Par; Mylan; Valeant

SUMMARY:
Determine bioequivalence between branded and generic bupropion extended release (XL) products (and between generic products) at steady state in patients with major depressive disorder.

DETAILED DESCRIPTION:
The protocol is a prospective, randomized, double-blinded, crossover study with Major Depressive Disorder (MDD) receiving bupropion HCl 300mg XL (branded or generic).

Subjects will be studied in 4 phases for a total of approximately 28 weeks:

Phase 1: an approximately 4-week lead-in phase during which participants remain on their existing bupropion product Phases 2 - 4: randomized cross-over phases of approximately 6 weeks on each of the four bupropion study drugs (brand and 3 generics).

ELIGIBILITY:
Inclusion Criteria

Each subject must meet all of the following criteria:

1. Adult outpatients age 18-75 years
2. Currently on once daily bupropion HCl 300mg XL (brand or any generic), for a minimum of 4 months
3. Major depressive disorder (MDD), in partial or full remission for at least 4 months, as confirmed by the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID). Spontaneous relapse of depression unrelated to medication changes is less likely - about 5% chance per year - after remission has been maintained for at least 4 months.2
4. Ability to understand and willingness to comply with study procedures, and to provide written informed consent

Exclusion Criteria

Subjects will not be enrolled if any of the following criteria exist:

1. Remission from depression not clearly attributed to bupropion treatment
2. Current severe side effects attributable to bupropion
3. Poor adherence to bupropion treatment per patient self- report and history of refill persistence
4. History of active seizure disorder, or seizure treatment within past year
5. History of significant hepatic or renal disease, based on physician assessment
6. Currently taking drugs or natural products known to influence cytochrome P450B6 (CYP2B6) activity
7. Currently taking drugs for hepatitis C or multiple sclerosis, due to their ability to cause depression
8. Dementia or other significant cognitive impairment, per diagnosis or investigative team's assessment
9. Lifetime diagnosis of schizophrenia, schizoaffective or schizophreniform dis-order, delusional disorder, or current psychotic symptoms diagnosed by SCID
10. Abuse of or dependence on alcohol or other substances within the past 6 months as determined by SCID, and confirmed by study physician interview
11. Current suicidal ideation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2014-06-25 (Actual); Primary Completion 2016-08-14 (Actual); Study Completion 2016-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evan D Kharasch, MD, PhD, Principal Investigator — Washington Univesity School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bupropion: Phase 1: (Non-randomized) an approximately 4-week lead-in phase during which participants remain on their existing bupropion product
  Other Names:
  Wellbutrin Par Mylan Valeant
Period: Phase 1 Current Tx (Non-randomized)
Arm/Group | Bupropion
Started | 74
Completed | 71
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 1
Period: Phase 2 (Randomized: 1 Brand, 3 Generic)
Arm/Group | Bupropion
Started | 71
Completed | 67
Not Completed | 4
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 1
Period: Phase 3 (Randomized: 1 Brand, 3 Generic)
Arm/Group | Bupropion
Started | 67
Completed | 67
Not Completed | 0
Period: Phase 4 (Randomized: 1 Brand, 3 Generic)
Arm/Group | Bupropion
Started | 67
Completed | 67
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Bupropion: Subjects will be studied for 28 weeks in a sequential cross-over study:
  1. a 4-week lead-in phase during which all participants remain on their existing bupropion product
  2. Four randomized cross-over phases of 6 weeks on each of the four bupropion study drugs (brand Wellbutrin 300mg XL, Valeant, Par and Watson 3 generics)
Arm/Group | Bupropion
Number analyzed (Participants) | 70
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 47 [37 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC0-24) Ratio for Racemic Bupropion
Description: Area under the curve (AUC) generic/Area under the curve (AUC) brand bupropion
Time Frame: For 24 hours approximately every 6 weeks
Measure: Mean (Full Range); unit: percentage of Brand
Groups:
- Valeant Brand Bupropion XL® 300mg; Par Generic Bupropion XL® 300mg; Watson Generic Bupropion XL® 300mg; Mylan Generic Bupropion XL® 300mg: Phase 1: an approximately 4-week lead-in phase during which participants remain on their existing bupropion product Phases 2 - 4: randomized cross-over phases of approximately 6 weeks on each of the four bupropion study drugs (brand and 3 generics).
Arm/Group | Valeant Brand Bupropion XL® 300mg | Par Generic Bupropion XL® 300mg | Watson Generic Bupropion XL® 300mg | Mylan Generic Bupropion XL® 300mg
Number analyzed (Participants) | 67 | 67 | 67 | 67
percentage of Brand
  Bupropion | .84 [.71 to 1.04] | .88 [.72 to 1.08] | .83 [.68 to .99] | .89 [.7 to 1.06]
  Hydroxybupropion | 20.9 [15.5 to 25.5] | 20.9 [15.9 to 28.1] | 21.8 [15.9 to 26.5] | 21.6 [15.9 to 27.7]
  Erthrohydrobuprion | 2.09 [1.52 to 2.59] | 2.05 [1.47 to 2.57] | 1.98 [1.48 to 2.34] | 2.02 [1.61 to 2.50]
  Threohydrobupropion | 9.38 [7.21 to 13.27] | 9.05 [7.21 to 13.27] | 8.57 [6.83 to 11.57] | 8.78 [7.25 to 12.49]
Statistical Analysis 1: Comparison: Valeant Brand Bupropion XL® 300mg vs Par Generic Bupropion XL® 300mg vs Watson Generic Bupropion XL® 300mg vs Mylan Generic Bupropion XL® 300mg; Test type: Superiority; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: 28 weeks
Arm/Group | Valeant Brand Bupropion XL® 300mg | PAR Generic Bupropion XL® 300mg | Watson Generic Bupropion XL® 300mg | Mylan Generic Bupropion XL® 300mg
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/71 | 0/71 | 0/71
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/71 | 0/71 | 0/71
Other Adverse Events (participants affected / at risk) | 0/71 | 0/71 | 1/71 | 0/71
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valeant Brand Bupropion XL® 300mg (N=71) | PAR Generic Bupropion XL® 300mg (N=71) | Watson Generic Bupropion XL® 300mg (N=71) | Mylan Generic Bupropion XL® 300mg (N=71)
depression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-19): https://cdn.clinicaltrials.gov/large-docs/97/NCT02209597/Prot_SAP_000.pdf